CLINICAL TRIAL: NCT00197587
Title: Prevention of Milk-Borne Transmission of HIV-1C in Botswana ("Mashi")
Brief Title: Prevention of Milk-Borne Transmission of HIV-1C in Botswana
Acronym: Mashi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Max Essex, Study Chair, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HSC 10411/9912BOTS
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infection; Infant Risk for HIV Infection by MTCT
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- maternal nevirapine (Active Comparator)
  Interventions: Drug: Nevirapine
- maternal placebo (Placebo Comparator)
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: Nevirapine — All women received a background of zidovudine from 34 weeks' gestation through delivery, and all infants received single-dose nevirapine at birth and zidovudine from birth through 1 month. Women were randomized to receive either single-dose nevirapine or placebo during labor.
  Arms: maternal nevirapine
Drug: No intervention — All women received a background of zidovudine from 34 weeks'gestation through delivery, and all infants received single-dose nevirapine at birth and zidovudine from birth through 1 month. Women were randomized to receive either single-dose nevirapine or placebo during labor.
  Arms: maternal placebo

SUMMARY:
The purpose of this study is to find the most effective and safe treatment to prevent the passage of HIV from an infected mother to her baby.

DETAILED DESCRIPTION:
1. To assess the effectiveness of the addition of a single dose of nevirapine (NVP) to Zidovudine (ZDV, also known as AZT) as used in the Botswana mother-to-child transmission (MTCT) National Program, in reducing transmission of HIV-1 from mother to child. To determine if maternal NVP (per HIVNET 012 protocol) is necessary in the setting of maternal ZDV from 34 weeks gestation through delivery AND single-dose prophylactic infant NVP at birth plus ZDV from birth to 4 weeks for the reduction of transmission of HIV-1 from mother to child.
2. To assess the effect of prophylactic AZT given to infants during breast feeding on HIV transmission.
3. To confirm the safety and tolerance of one dose of NVP given to mothers and infants
4. To evaluate the safety and tolerance of AZT given to infants for up to 6 months of age
5. To determine the association between assigned infant feeding strategy and maternal morbidity and mortality
6. To determine the rates of virologic response to NNRTI-containing HAART at 26 and 52 weeks after initiating treatment, among HIV+ women who previously received single dose NVP versus placebo during labour.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must be no more than 34 weeks pregnant, intending to carry to term, intending to stay in area for at least 7 months, and consenting to HIV-1 testing and participation; HIV-1 infected by ELISA confirmed by Western blot; etc.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2002-08; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
HIV PCR | 1 month
  The primary endpoint was infant HIV infection by the
  1-month visit.

CONTACTS AND LOCATIONS:
Overall Officials: Myron Essex, DVM,PhD, Study Chair — Harvard School of Public Health (HSPH)

REFERENCES:
- [Result] Thior I, Lockman S, Smeaton LM, Shapiro RL, Wester C, Heymann SJ, Gilbert PB, Stevens L, Peter T, Kim S, van Widenfelt E, Moffat C, Ndase P, Arimi P, Kebaabetswe P, Mazonde P, Makhema J, McIntosh K, Novitsky V, Lee TH, Marlink R, Lagakos S, Essex M; Mashi Study Team. Breastfeeding plus infant zidovudine prophylaxis for 6 months vs formula feeding plus infant zidovudine for 1 month to reduce mother-to-child HIV transmission in Botswana: a randomized trial: the Mashi Study. JAMA. 2006 Aug 16;296(7):794-805. doi: 10.1001/jama.296.7.794. PMID 16905785
- [Result] Shapiro RL, Thior I, Gilbert PB, Lockman S, Wester C, Smeaton LM, Stevens L, Heymann SJ, Ndung'u T, Gaseitsiwe S, Novitsky V, Makhema J, Lagakos S, Essex M. Maternal single-dose nevirapine versus placebo as part of an antiretroviral strategy to prevent mother-to-child HIV transmission in Botswana. AIDS. 2006 Jun 12;20(9):1281-8. doi: 10.1097/01.aids.0000232236.26630.35. PMID 16816557
- [Result] Lockman S, Shapiro RL, Smeaton LM, Wester C, Thior I, Stevens L, Chand F, Makhema J, Moffat C, Asmelash A, Ndase P, Arimi P, van Widenfelt E, Mazhani L, Novitsky V, Lagakos S, Essex M. Response to antiretroviral therapy after a single, peripartum dose of nevirapine. N Engl J Med. 2007 Jan 11;356(2):135-47. doi: 10.1056/NEJMoa062876. PMID 17215531
- [Derived] Powis KM, Smeaton L, Hughes MD, Tumbare EA, Souda S, Jao J, Wirth KE, Makhema J, Lockman S, Fawzi W, Essex M, Shapiro RL. In-utero triple antiretroviral exposure associated with decreased growth among HIV-exposed uninfected infants in Botswana. AIDS. 2016 Jan;30(2):211-20. doi: 10.1097/QAD.0000000000000895. PMID 26684818
- [Derived] Dryden-Peterson S, Jayeoba O, Hughes MD, Jibril H, McIntosh K, Modise TA, Asmelash A, Powis KM, Essex M, Shapiro RL, Lockman S. Cotrimoxazole prophylaxis and risk of severe anemia or severe neutropenia in HAART-exposed, HIV-uninfected infants. PLoS One. 2013 Sep 23;8(9):e74171. doi: 10.1371/journal.pone.0074171. eCollection 2013. PMID 24086319
- [Derived] Dryden-Peterson S, Shapiro RL, Hughes MD, Powis K, Ogwu A, Moffat C, Moyo S, Makhema J, Essex M, Lockman S. Increased risk of severe infant anemia after exposure to maternal HAART, Botswana. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):428-36. doi: 10.1097/QAI.0b013e31820bd2b6. PMID 21266910
- [Derived] Powis KM, Smeaton L, Ogwu A, Lockman S, Dryden-Peterson S, van Widenfelt E, Leidner J, Makhema J, Essex M, Shapiro RL. Effects of in utero antiretroviral exposure on longitudinal growth of HIV-exposed uninfected infants in Botswana. J Acquir Immune Defic Syndr. 2011 Feb 1;56(2):131-8. doi: 10.1097/QAI.0b013e3181ffa4f5. PMID 21124227